CLINICAL TRIAL: NCT01427647
Title: Inflammatory Response Following Colorectal Cancer Surgery Depends on the Type of Anesthesia and Surgery
Brief Title: Inflammatory Response After Colorectal Cancer Surgery
Acronym: CRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Patricia Duque, M.D., Anesthesiologist staff, Universidad Complutense de Madrid
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Complutense University 1
Record Dates: First submitted 2011-08-29; First posted 2011-09-01 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer
Keywords: Laparoscopy; Anesthesia, Epidural
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (Active Comparator): Control group: open surgery under general anesthesia
  Interventions: Procedure: Laparoscopic technique and thoracic epidural anesthesia
- Epidural group (Active Comparator): Epidural group: Open surgery under thoracic epidural anesthesia
  Interventions: Procedure: Laparoscopic technique and thoracic epidural anesthesia
- Laparoscopic group (Active Comparator): Laparoscopic group: Laparoscopic surgery under general anesthesia
  Interventions: Procedure: Laparoscopic technique and thoracic epidural anesthesia

INTERVENTIONS:
Procedure: Laparoscopic technique and thoracic epidural anesthesia — We have compared colorectal cancer surgery under two types of surgical(laparoscopic versus open) and anesthesia (thoracic epidural versus general) techniques

SUMMARY:
Laparoscopic technique and epidural anesthesia have been proposed to improve postoperative outcome following colorectal cancer surgery. The investigators hypothesize that the inflammatory response is attenuated by laparoscopic surgery and epidural anesthesia compared to traditional open surgery under general anesthesia.

DETAILED DESCRIPTION:
Patients scheduled for open colorectal cancer surgery were randomly allocated to receive general anesthesia (CON group, n=22) or general anesthesia with thoracic epidural anesthesia (EPI group, n=21). Patients undergoing laparoscopic surgery (LAP group, n=20) composed the third arm of the study. Measurement of perioperative changes in several hormones and cytokines were blinded to group assignment.

Primary outcome: Compare simultaneously two types of surgical and anesthesia techniques for colorectal cancer surgery and measure to what extent the stress response is lessened.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for colorectal cancer surgery

Exclusion Criteria:

* Emergent surgery
* Intestinal obstruction
* Contraindication for epidural catheter placement
* Concomitant autoimmune disease
* Concomitant infectious disease
* Recent corticosteroids or anti-inflammatory medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2007-06; Primary Completion 2009-05 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Plasma levels of several cytokines after colorectal cancer surgery | within the first two days after surgery
  We have measured and compared perioperative plasma levels of interleukin-1, interleukin-2, interleukin-6,monocyte chemotactic protein-1, interleukin-8, nitric oxide, C-reactive protein and procalcitonin in our three-group sample.

SECONDARY OUTCOMES:
Incidence of adverse clinical outcomes between groups | within 30 days after surgery
  We have analyzed if there is any significant difference on respiratory, cardiac, renal or infectious postoperative complications between groups

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Duque, MD, Principal Investigator — Gregorio Marañon Hospital
Locations (1):
- Gregorio Marañon Hospital, Madrid, Madrid, Spain